CLINICAL TRIAL: NCT03994510
Title: Study of Shame Propensity as a Prognostic Factor of Suicidal Behaviors in Patients With Borderline Personality Disorder
Brief Title: SHame prOpensity in bOrderline Personality Disorder
Acronym: SHOO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM 1061, " Neuropsychiatry: epidemiological and clinical research", Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0286
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Borderline Personality Disorder
Keywords: Psychiatry; Suicidal Behavior; Borderline Personality Disorder; Follow-Up Study
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: During each visit, a clinical evaluation will be carried out, as well as the filling of hetero-questionnaires and self-questionnaires. Two biological collections will be made: one during the inclusion visit, and the other during the last visit, 5 years after inclusion.
  First visit (Baseline) only: Sociodemographic data, Clinical evaluation, family history
  At Baseline and 5 years after baseline only:
  * Blood sample
  * BPD diagnosis (using the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM) Disorders (SCID II))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Borderline Personality Disorder (Other): At each visit, these patients will have an interview that will allow for a clinical evaluation, as well as completing the hetero-questionnaires and self-questionnaires
  Interventions: Other: Clinical and biological assessments - a 5 Years follow-up

INTERVENTIONS:
Other: Clinical and biological assessments - a 5 Years follow-up — During each visit, a clinical evaluation will be carried out, as well as the filling of hetero-questionnaires and self-questionnaires. Two biological collections will be made: one during the inclusion visit, and the other during the last visit, 5 years after inclusion.

SUMMARY:
Borderline Personality Disorder (BPD) is a common psychiatric disorder occurring in 2 to 6% of the population. 70% of patients with BPD do at least one Suicide Attempt (SA) in their lives. It makes BPD the most related to SA condition.

Negative interpersonal events are among the main stressor inducing a SA. Patients with BPD are characterized by emotional dysregulation, impulsivity (repeated parasuicidal and suicidal behaviors), and instability in interpersonal relationships. The feeling of shame related to this psychiatric disorder could be one of the causes of the high SA rate. In this study, patients with BPD will be follow-up during 5 years.

The main objective is to study the propensity to feel shame as a predictor of SA.

This include:

* Study of shame propensity as a predictive factor of suicidal behavior - Identify homogeneous subgroups of patients with BPD based on SA, and overall functioning.
* Identify biological markers predicting SA
* Identify predictive and protective treatments (pharmacological and psychotherapeutic) for SA

DETAILED DESCRIPTION:
This is a 5 years follow-up prospective study recruiting 688 patients.

Schedule of the study :

Inclusion period : 3 years Duration of follow-up of each patient : 5 years Estimated duration of the study : 8.5 years

As part of the research, patients will be summoned annually for 5 years.

The first visit (at baseline) is included in the usual care

The follow-up visits are specifics to the research

During the visits patients will complete self questionary and clinical interview.

The organization of visits is as follows:

* an inclusion visit lasting around 2 hours (clinical evaluation and then self-questionnaires)
* a visit to 1 year, 2 years, 3 years, 4 years and 5 years (+/- 1 month) lasting approximately 1 hour 30 (clinical evaluation and passing of self-questionnaires)

Genetic samples will be taken during the initial visit as well as during the visit to 5 years.

They consist of:

* A genetic collection consisting of a DNA library (3 Ethylene Diamine Triacetic Acid (EDTA) tubes of 6ml - 18 ml).
* An off-genetics collection consisting of serum and plasma samples, (1 6 ml EDTA tube, 1 4 ml heparinized tube, 2 dry tubes of 5 ml each and 2 citrated tubes of 2.7 ml each - 25 , 4 ml).

ELIGIBILITY:
Inclusion criteria:

* To be over 18
* Clinical diagnosis of BPD using the SCID II (Structured Clinical Interview for DSM-IV-Text Reviewed Axis II Personality Disorders)
* Having signed the informed consent
* Able to understand the nature, the purpose and the methodology of the study
* Able to understand and perform the clinical evaluations

Exclusion criteria:

* Deprived of liberty (by judicial or administrative decision)
* Protected by law (guardianship)
* Exclusion period in relation to another protocol
* Not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Level of shame propensity | At enrollment
  Evaluation of the level of shame propensity will be measured using the Test of Self Conscious Affect (TOSCA)
Level of shame propensity | 1 year after enrollment
  Evaluation of the level of shame propensity will be measured using the Test of Self Conscious Affect (TOSCA)
Level of shame propensity | 2 years after enrollment
  Evaluation of the level of shame propensity will be measured using the Test of Self Conscious Affect (TOSCA)
Level of shame propensity | 3 years after enrollment
  Evaluation of the level of shame propensity will be measured using the Test of Self Conscious Affect (TOSCA)
Level of shame propensity | 4 years after enrollment
  Evaluation of the level of shame propensity will be measured using the Test of Self Conscious Affect (TOSCA)
Level of shame propensity | 5 years after enrollment
  Evaluation of the level of shame propensity will be measured using the Test of Self Conscious Affect (TOSCA)
Number of SA compared to the clinical data obtained in baseline | At enrollment
  The number of SA will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the clinical data obtained in baseline
Number of SA compared to the clinical data obtained in baseline | 1 year after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the clinical data obtained in baseline
Number of SA compared to the clinical data obtained in baseline | 2 years after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the clinical data obtained in baseline
Number of SA compared to the clinical data obtained in baseline | 3 years after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the clinical data obtained in baseline
Number of SA compared to the clinical data obtained in baseline | 4 years after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the clinical data obtained in baseline
Number of SA compared to the clinical data obtained in baseline | 5 years after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the clinical data obtained in baseline

SECONDARY OUTCOMES:
Number of SA compared to the biological data obtained in baseline | At enrollment
  The number of SA will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the biological data obtained in baseline
Number of SA compared to the biological data obtained in baseline | 1 year after enrollment
  The number of SA will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the biological data obtained in baseline
Number of SA compared to the biological data obtained in baseline | 2 years after enrollment
  The number of SA will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the biological data obtained in baseline
Number of SA compared to the biological data obtained in baseline | 3 years after enrollment
  The number of SA will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the biological data obtained in baseline
Number of SA compared to the biological data obtained in baseline | 4 years after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the biological data obtained in baseline
Number of SA compared to the biological data obtained in baseline | 5 years after enrollment
  The number of SA within the year will be collected using Columbia Suicide Severity Rating Scale (C-SSRS) and compared to the biological data obtained in baseline
Suicidal Ideation | At enrollment
  The number of suicidal ideation will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Suicidal Ideation | 1 year after enrollment
  The number of suicidal ideation will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Suicidal Ideation | 2 years after enrollment
  The number of suicidal ideation will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Suicidal Ideation | 3 years after enrollment
  The number of suicidal ideation will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Suicidal Ideation | 4 years after enrollment
  The number of suicidal ideation will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Suicidal Ideation | 5 years after enrollment
  The number of suicidal ideation will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Parasuicidal Behaviours | At enrollment
  The number of parasuicidal behaviours will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Parasuicidal Behaviours | 1 year after enrollment
  The number of parasuicidal behaviours will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Parasuicidal Behaviours | 2 years after enrollment
  The number of parasuicidal behaviours will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Parasuicidal Behaviours | 3 years after enrollment
  The number of parasuicidal behaviours will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Parasuicidal Behaviours | 4 years after enrollment
  The number of parasuicidal behaviours will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Parasuicidal Behaviours | 5 years after enrollment
  The number of parasuicidal behaviours will be collected using Columbia Suicide Severity Rating Scale (C-SSRS).
Sick leave for a psychiatric condition | At enrollment
  The number of sick leaves, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Sick leave for a psychiatric condition | 1 year after enrollment
  The number of sick leaves, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Sick leave for a psychiatric condition | 2 years after enrollment
  The number of sick leaves, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Sick leave for a psychiatric condition | 3 years after enrollment
  The number of sick leaves, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Sick leave for a psychiatric condition | 4 years after enrollment
  The number of sick leaves, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Sick leave for a psychiatric condition | 5 years after enrollment
  The number of sick leaves, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Hospitalization for a psychiatric condition | At enrollment
  The number of hospitalization, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Hospitalization for a psychiatric condition | 1 year after enrollment
  The number of hospitalization, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Hospitalization for a psychiatric condition | 2 years after enrollment
  The number of hospitalization, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Hospitalization for a psychiatric condition | 3 years after enrollment
  The number of hospitalization, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Hospitalization for a psychiatric condition | 4 years after enrollment
  The number of hospitalization, related to BPD, and their duration will be collected and reported on the case report form (CRF).
Hospitalization for a psychiatric condition | 5 years after enrollment
  The number of hospitalization, related to BPD, and their duration will be collected and reported on the case report form (CRF).
The need to emergency psychiatric consult | At enrollment
  The number of emergency visit related to BPD, will be collected and reported on the case report form (CRF).
The need to emergency psychiatric consult | 1 year after enrollment
  The number of emergency visit related to BPD, will be collected and reported on the case report form (CRF).
The need to emergency psychiatric consult | 2 years after enrollment
  The number of emergency visit related to BPD, will be collected and reported on the case report form (CRF).
The need to emergency psychiatric consult | 3 years after enrollment
  The number of emergency visit related to BPD, will be collected and reported on the case report form (CRF).
The need to emergency psychiatric consult | 4 years after enrollment
  The number of emergency visit related to BPD, will be collected and reported on the case report form (CRF).
The need to emergency psychiatric consult | 5 years after enrollment
  The number of emergency visit related to BPD, will be collected and reported on the case report form (CRF).
Major depressive episodes | At enrollment
  The number of major depressives episodes and the measure of the depression intensity will be collected using the Inventory of Depressive Symptomatology (IDS-C30).
Major depressive episodes | 1 year after enrollment
  The number of major depressives episodes and the measure of the depression intensity will be collected using the Inventory of Depressive Symptomatology (IDS-C30).
Major depressive episodes | 2 years after enrollment
  The number of major depressives episodes and the measure of the depression intensity will be collected using the Inventory of Depressive Symptomatology (IDS-C30).
Major depressive episodes | 3 years after enrollment
  The number of major depressives episodes and the measure of the depression intensity will be collected using the Inventory of Depressive Symptomatology (IDS-C30).
Major depressive episodes | 4 years after enrollment
  The number of major depressives episodes and the measure of the depression intensity will be collected using the Inventory of Depressive Symptomatology (IDS-C30).
Major depressive episodes | 5 years after enrollment
  The number of major depressives episodes and the measure of the depression intensity will be collected using the Inventory of Depressive Symptomatology (IDS-C30).
Global functioning | At enrollment
  The Global functioning will be measured using the Functioning Assessment Short Test (FAST).
Global functioning | 1 year after enrollment
  The Global functioning will be measured using the Functioning Assessment Short Test (FAST).
Global functioning | 2 years after enrollment
  The Global functioning will be measured using the Functioning Assessment Short Test (FAST).
Global functioning | 3 years after enrollment
  The Global functioning will be measured using the Functioning Assessment Short Test (FAST).
Global functioning | 4 years after enrollment
  The Global functioning will be measured using the Functioning Assessment Short Test (FAST).
Global functioning | 5 years after enrollment
  The Global functioning will be measured using the Functioning Assessment Short Test (FAST).
Life Quality | At enrollment
  The Life Quality will be measured using the Satisfaction With Life Scale (SWLS).
Life Quality | 1 year after enrollment
  The Life Quality will be measured using the Satisfaction With Life Scale (SWLS).
Life Quality | 2 years after enrollment
  The Life Quality will be measured using the Satisfaction With Life Scale (SWLS).
Life Quality | 3 years after enrollment
  The Life Quality will be measured using the Satisfaction With Life Scale (SWLS).
Life Quality | 4 years after enrollment
  The Life Quality will be measured using the Satisfaction With Life Scale (SWLS).
Life Quality | 5 years after enrollment
  The Life Quality will be measured using the Satisfaction With Life Scale (SWLS).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No